CLINICAL TRIAL: NCT03393949
Title: Effect of Preoperative Low-dose of Methylprednisolone on Postoperative Pain and Immune Functions After Video-assisted Thoracoscopic Surgery: A Prospective Randomized Controlled Trial
Brief Title: Effects of Methylprednisolone on Immunological Function and Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, resident doctor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Effects of methylprednisolone
Record Dates: First submitted 2016-12-19; First posted 2018-01-09 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Methylprednisolone; Immunological Function; Postoperative Pain
Keywords: Methylprednisolone; Postoperative pain; Immunological function
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group M (Experimental): Patients in Group M received methylprednisolone 1mg•kg-1
  Interventions: Drug: Methylprednisolone 1 mg•kg-1
- Group C (Experimental): Patients in Group C received isotonic saline 1mg•kg-1
  Interventions: Drug: isotonic saline 1mg•kg-1

INTERVENTIONS:
Drug: Methylprednisolone 1 mg•kg-1 — Patients in Group M received methylprednisolone 1mg•kg-1
  Arms: Group M
Drug: isotonic saline 1mg•kg-1 — Patients in Group C received isotonic saline 1mg•kg-1
  Arms: Group C

SUMMARY:
Surgical trauma is characterized by a tightly integrated sequence of neurohumoral and immunological processes. When this is marked, it can manifest as a clinical entity called the systemic inflammatory response syndrome. Previous studies reported that inflammatory milieu in the postoperative period can be a harmful and potentially modifiable condition that may affect postoperative recovery, which includes the level of pain, fatigue, dizziness, nausea and vomiting (PONV), muscle weakness, and sleep quality and then increases the need for hospitalization. The effect of postoperative inflammation-related immune suppression such as the T-cell exhaustion and lymphocyte anergy may render the patient vulnerable to both infection and the recurrence of malignancy on postoperative infection risk and malignancy recurrence are currently subjects of intense speculation and investigation.

Glucocorticoids are well known for their analgesic, anti-inflammatory, immunosuppressive agents and antiemetic effects. Though previous studies' results on postoperative outcome have been positive and in favor of glucocorticoid use, with postoperative nausea and vomiting and pain outcome parameters most significantly improved. However, high-dose methylprednisolone treatment could result in decreases T-cells postoperatively. Based on these consideration, the aim of our study was to assess the effect of a single low-dose preoperative methylprednisolone (MP) 1 mg/Kg i.v. on postoperative pain and immune functions in patients undergoing video-assisted thoracoscopic surgery (VATS) under general anesthesia.

DETAILED DESCRIPTION:
The eighty-one patients were randomly assigned either to the MP Group or the Control Group in a 1:1 ratio using a computer-generated randomization number sequence. The group assignment was sealed in sequentially numbered opaque envelopes. No stratiﬁcation or block randomization was made. The envelopes were opened on the morning of surgery, and the trial drug was prepared by a senior anaesthetist not otherwise involved in data collection. The MP group received a single-dose of MP, 1 mg/Kg i.v. (Solu-Medrolw; Pﬁzer, Ballerup, Denmark) and the Control group a single-dose of isotonic saline ( equal capacity with MP) i.v. The test solution was administered just 30 mins before the operation. The patients, attending anesthesiologists, surgeons, and data collectors were all blinded to patient group assignment.The primary outcomes of the levels of T lymphocyte subsets of CD3+, CD4+, and CD8+, and the CD4+/CD8+ ratio were measured at T0, T1, and T2. Postoperative pain scores were evaluated by the visual analog scale (VAS) score16, where 0 indicates painlessness, and 10 indicates severe pain. The patients were asked to evaluate their pain at rest and during coughing at 2, 4, 6, and 24 hours postoperatively. Total pump press numbers of PCA and adverse effects during 24 hours after surgery such as hypotension, bradycardia, nausea and vomiting, and dizzy were recorded and treated accordingly.

ELIGIBILITY:
Inclusion Criteria:

* ASA Ⅱ～Ⅲ
* aged 65-85years
* consciousness,with no psychological or communication disorders, with educational level above primary school (including primary school).
* with no chemotherapy or radiotherapy before admission.
* no history of medicine allergy.
* no evident abnormality of liver, kidney or nervous system
* scheduled for radical operation for lung cancer under general anesthesia

Exclusion Criteria:

* diagnosed with diseases in nervous system or psychological disorder, history of taking sedatives or anti-depressants.
* history of hypertension, diabetes, coronary heart disease, cerebral infarction.
* had drugs which affect immunological function before.
* severe acuity or vision dysfunction or have difficulty in communication.
* with special complications during surgery.
* had blood transfusion treatment during perioperation period history of heart operation
* Mini-mental State Examination Scores less than 25 before surgery.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Change in the level of T lymphocyte subsets cluster of differentiation 3(CD3+) | Baseline, the end of surgery, 24 hours after surgery
  Tested the level of CD3+ with flow cytometry at the time points of pre-induction (T0), the end of surgery (T1) and 24h after surgery (T2)
Change in the level of T lymphocyte subsets cluster of differentiation 4(CD4+) | Baseline, the end of surgery, 24 hours after surgery
  Tested the level of CD4+ with flow cytometry at the time points of pre-induction (T0), the end of surgery (T1) and 24h after surgery (T2)
Change in the level of T lymphocyte subsets cluster of differentiation 8(CD8+) | Baseline, the end of surgery, 24 hours after surgery
  Tested the level of CD4+ with flow cytometry at the time points of pre-induction (T0), the end of surgery (T1) and 24h after surgery (T2)
The ratio of T lymphocyte subsets cluster of differentiation 4(CD4+)/ T lymphocyte subsets cluster of differentiation 8(CD8+) | Baseline, the end of surgery, 24 hours after surgery
  Calculated the ratio of CD4+/CD8+ at the time points of pre-induction (T0), the end of surgery (T1) and 24h after surgery (T2)

SECONDARY OUTCOMES:
postoperative pain score | 2, 4 6, 24 hours after surgery
  Tested postoperative pain by using visual analog scale
Adverse effect | 24 hours after surgery
  Tested postoperative adverse effect

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Zhu, doctor, Study Director — professor
Locations (1):
- Shengjing hospital of China medical university, Shenyang, Liaoning, China